CLINICAL TRIAL: NCT05435599
Title: Efficacy of Serum Regucalcin Level in Detecting Fibrosis in Chronic Hepatitis B Infection
Brief Title: Serum Regucalcin Level and Chronic Hepatitis B
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konya Meram State Hospital (Other)
Responsible Party: Principal Investigator, Fatma Çölkesen, Principal Investigator, Konya Meram State Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 10542
Record Dates: First submitted 2021-12-06; First posted 2022-06-28 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Chronic Hepatitis b; Liver Fibrosis
Keywords: hepatitis b; fibrosis; regucalcin; liver
MeSH Terms: conditions — Hepatitis B, Chronic; Liver Cirrhosis; Hepatitis B; Fibrosis

STUDY DESIGN:
Intervention Model Description: Patients undergoing liver biopsy for chronic hepatitis b
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chronic Hepatitis B (Other): Measurement of serum regucalcin level
  Interventions: Diagnostic Test: Serum regucalcin level
- Healthy Volunteers (Other): Measurement of serum regucalcin level
  Interventions: Diagnostic Test: Serum regucalcin level

INTERVENTIONS:
Diagnostic Test: Serum regucalcin level — During routine outpatient controls, serum regucalcin level will be measured from the rest of the blood taken for examinations.

SUMMARY:
This study, it was aimed to investigate the relationship between serum regucalcin level and liver fibrosis level in patients with CHB infection.

DETAILED DESCRIPTION:
Chronic hepatitis B (CHB) infection continues to be an important health problem due to its high morbidity and mortality. For this reason, it is very important to determine the appropriate timing to start antiviral therapy in patients with CHB infection and to evaluate the stage of liver fibrosis in the treatment follow-up. Liver biopsy is the gold standard for detecting liver fibrosis. Although it is generally accepted to be a safe procedure, it can cause some serious complications. For this reason, in recent years, many studies have been conducted on new noninvasive tests in the evaluation of liver fibrosis. One of them is the serum regucalcin level. Studies have shown that serum regucalcin levels increase in liver damage, but there is no study in the literature comparing liver fibrosis and serum regucalcin levels in CHB infection. This study, it was aimed to investigate the relationship between serum regucalcin level and liver fibrosis level in patients with CHB infection.

ELIGIBILITY:
Inclusion Criteria:

* Being followed up with a diagnosis of chronic hepatitis B
* Not having a known history of liver disease who applied to our outpatient clinic for other reasons
* Having a liver biopsy
* ≥18 years

Exclusion Criteria:

* <18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Comparison of serum regucalcin levels with liver fibrosis levels | Performing liver biopsies: 3 months, data collection: 1 month, writing the article: 1 month
  We grouped chronic hepatitis b patients as mild fibrosis (stage 1-2) and moderate fibrosis (stage 3-4) according to the fibrosis stage at liver biopsy stage. We selected healthy volunteers without liver disease as the control group. We will measure the serum regucalcin level in these 3 groups and make a comparison between the groups. We want to show the relationship between serum regucalcin level and fibrosis level in chronic hepatitis b.

CONTACTS AND LOCATIONS:
Locations (1):
- Konya Training and Research Hospital, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wei X, Yu H, Zhao P, Xie L, Li L, Zhang J. Serum regucalcin is a useful indicator of liver injury severity in patients with hepatitis B virus-related liver diseases. Braz J Med Biol Res. 2019 Sep 30;52(10):e8845. doi: 10.1590/1414-431X20198845. eCollection 2019. PMID 31576907
- [Background] Yamaguchi M, Isogai M, Shimada N. Potential sensitivity of hepatic specific protein regucalcin as a marker of chronic liver injury. Mol Cell Biochem. 1997 Feb;167(1-2):187-90. doi: 10.1023/a:1006859121897. PMID 9059996